CLINICAL TRIAL: NCT05062889
Title: Exploiting Circulating Tumour DNA to Intensify the Postoperative Treatment of Stage III and High-risk Stage II Resected Colon Cancer Patients With Adjuvant FOLFOXIRI and/or Post-adjuvant Trifluridine/Tipiracil
Brief Title: Exploiting Circulating Tumour DNA to Intensify the Postoperative Treatment Resected Colon Cancer Patients
Acronym: ERASE-CRC
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: due to earlier termination of the agreement between the Sponsor and Central Laboratory for screening test. Enrollment will reopen as soon as a new laboratory is identified.
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Servier (Industry); Foundation Medicine (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERASE-CRC
Record Dates: First submitted 2021-09-13; First posted 2021-09-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Stage II Colon Cancer; Stage III Colon Cancer; HER2-positive Colon Cancer; RAS Wild-type Colon Cancer
Keywords: Circulating tumor DNA; FOLFOX; CAPOX; FOLFOXIRI; Trifluridine/Tipiracil; Trastuzumab; Tucatinib
MeSH Terms: conditions — Colonic Neoplasms | interventions — Fluorouracil; Leucovorin; Capecitabine; Irinotecan; trifluridine tipiracil drug combination; Trastuzumab; tucatinib

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, multicentre study, including two phase II randomized trials (Part 1 and Part 2) and a non-randomized cohort (Part 1 target-driven)
  In Part 1 resected stage III and high-risk stage II colon cancer patients with positive ct- DNA after surgery will be randomized to receive FOLFOX for 12 cycles or CAPOX for 8 cycles (at investigator choice) versus FOLFOXIRI for 12 cycles;
  In Part 1 target-driven resected stage III and high-risk stage II HER2+ RAS wild-type colon cancer patients with positive ct-DNA after surgery will receive Trastuzumab and Tucatinib plus FOLFOX for 12 cycles.
  In Part 2 resected stage III and high-risk stage II colon cancer patients with positive ct- DNA after the end of a fluoropyrimidine and oxaliplatin-based adjuvant therapy - either in the frame or outside of Part 1 - will be randomized to receive observation or Trifluridine/Tipiracil for 6 cycles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm B FOLFOXIRI, part 1 (adjuvant) (Experimental): FOLFOXIRI Irinotecan 165 mg/sqm iv over 60 minutes day 1, followed by Oxaliplatin 85 mg/sqm iv over 2 hours day 1, in two-way with L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 followed by 5-fluoruracil 3200 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. In the case of oxaliplatin and/or irinotecan interruption because of adverse events, patient's refusal or investigator's choice, the continuation of the other drugs until 12 cycles is recommended.
  Interventions: Drug: 5-Fluorouracil continuous infusion FOLFOXIRI schedule; Drug: Oxaliplatin FOLFOX and FOLFOXIRI schedule; Drug: L-Leucovorin; Drug: Irinotecan
- Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant) (Active Comparator): mFOLFOX6 Oxaliplatin 85 mg/sqm iv over 2 hours, day 1 in two-way with L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 followed by 5-fluorouracil 400 mg/sqm iv bolus, day 1 followed by 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. The continuation of 5FU/leucovorin until 12 cycles is recommended also if oxaliplatin is interrupted because of adverse events, patient's refusal or investigator's choice.
  CAPOX Oxaliplatin 130 mg/sqm iv over 2 hours, day 1; Capecitabine 1000 mg/sqm/bid per os from day 1 to day 14; to be repeated every 3 weeks until 8 cycles. The continuation of Capecitabine until 8 cycles is recommended also if oxaliplatin is interrupted because of adverse events, patient's refusal or investigator's choice.
  Pending the results of ct-DNA analysis, up to 2 cycles of FOLFOX/CAPOX before randomization are allowed to start the adjuvant treatment within 8-10 weeks after surgery
  Interventions: Drug: 5-Fluorouracil bolus FOLFOX schedule; Drug: 5-Fluorouracil continuous infusion FOLFOX schedule; Drug: Oxaliplatin FOLFOX and FOLFOXIRI schedule; Drug: Oxaliplatin CAPOX schedule; Drug: L-Leucovorin; Drug: Capecitabine
- Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant) (Experimental): Tucatinib 300 mg (two 150 mg tablets)/bid orally twice daily (approximately 8 to 12 hours between doses with or without a meal); Trastuzumab 4 mg/kg iv over 30 minutes, day 1 (loading dose: 6 mg/kg iv over 90 minutes), followed by
  mFOLFOX6 Oxaliplatin 85 mg/sqm iv over 2 hours, day 1 in two-way with L-Leucovorin 200 mg/sqm iv over 2 hours, day 1 followed by 5-fluorouracil 400 mg/sqm iv bolus, day 1 followed by 5-fluoruracil 2400 mg/sqm 48 h-continuous infusion, starting on day 1; to be repeated every 2 weeks for a maximum of 12 cycles. In the case of oxaliplatin and/or trastuzumab and/or tucatinib interruption because of adverse events, patient's refusal or investigator's choice, the prosecution of the other drugs until 12 cycles is recommended.
  Pending the results of ct-DNA analysis, up to 2 cycles of FOLFOX/CAPOX before randomization are allowed to start the adjuvant treatment within 8-10 weeks after surgery
  Interventions: Drug: 5-Fluorouracil bolus FOLFOX schedule; Drug: 5-Fluorouracil continuous infusion FOLFOX schedule; Drug: Oxaliplatin FOLFOX and FOLFOXIRI schedule; Drug: Oxaliplatin CAPOX schedule; Drug: L-Leucovorin; Drug: Trastuzumab; Drug: Tucatinib
- Arm B Trifluridine/Tipiracil, part 2 (post-adjuvant) (Experimental): Trifluridine/Tipiracil: 35 mg/ m2/bid per os days 1-5 and 8-12 to be repeated every 4 weeks until 6 cycles.
  Interventions: Drug: Trifluridine/Tipiracil
- Arm A Observation, part 2 (post-adjuvant) (No Intervention): Follow-up

INTERVENTIONS:
Drug: 5-Fluorouracil continuous infusion FOLFOXIRI schedule — 3200 mg/sqm 48 h-continuous infusion, starting on day 1. To be repeated every two weeks for a maximum of 12 cycles.
  Other Names: 5FU
  Arms: Arm B FOLFOXIRI, part 1 (adjuvant)
Drug: 5-Fluorouracil bolus FOLFOX schedule — 400 mg/sqm iv bolus, day 1. To be repeated every two weeks for a maximum of 12 cycles.
  Other Names: 5FU
  Arms: Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant); Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)
Drug: 5-Fluorouracil continuous infusion FOLFOX schedule — 2400 mg/sqm 48 h-continuous infusion, starting on day 1. To be repeated every two weeks for a maximum of 12 cycles.
  Other Names: 5FU
  Arms: Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant); Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)
Drug: Oxaliplatin FOLFOX and FOLFOXIRI schedule — 85 mg/sqm iv over 2 hours, day 1. To be repeated every two weeks for a maximum of 12 cycles.
  Other Names: Oxa
  Arms: Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant); Arm B FOLFOXIRI, part 1 (adjuvant); Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)
Drug: Oxaliplatin CAPOX schedule — 130 mg/sqm iv over 2 hours, day 1. To be repeated every three weeks for a maximum of 8 cycles.
  Other Names: Oxa
  Arms: Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant); Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)
Drug: L-Leucovorin — 200 mg/sqm iv over 2 hours, day 1. To be repeated every two weeks for a maximum of 12 cycles.
  Other Names: Lederfolin
  Arms: Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant); Arm B FOLFOXIRI, part 1 (adjuvant); Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)
Drug: Capecitabine — Capecitabine 1000 mg/sqm/bid per os from day 1 to day 14. To be repeated every 3 weeks until 8 cycles. Available as 500 and 150 mg tablets.
  Arms: Arm A mFOLFOX6 or CAPOX (at investigator's choice), part 1 (adjuvant)
Drug: Irinotecan — 165 mg/sqm iv over 60 minutes, day 1. To be repeated every two weeks for a maximum of 12 cycles.
  Arms: Arm B FOLFOXIRI, part 1 (adjuvant)
Drug: Trifluridine/Tipiracil — 35 mg/m2/bid per os days 1-5 and 8-12. To be repeated every 4 weeks until 6 cycles. Available as 20 and 15 mg tablets.
  Other Names: FTD/TPI
  Arms: Arm B Trifluridine/Tipiracil, part 2 (post-adjuvant)
Drug: Trastuzumab — 4 mg/kg iv over 30 minutes, day 1 (loading dose: 6 mg/kg iv over 90 minutes). To be repeated every two weeks for a maximum of 12 cycles.
  Arms: Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)
Drug: Tucatinib — 300 mg (two 150 mg tablets)/bid orally twice daily (approximately 8 to 12 hours between doses with or without a meal) for a maximum of 12 biweekly cycles.
  Arms: Trastuzumab and Tucatinib plus mFOLFOX6, part 1 target-driven (adjuvant)

SUMMARY:
The aims of this study are to evaluate if an intensified adjuvant treatment with FOLFOXIRI could increase the rate of cases with undetectable ct-DNA after chemotherapy and to evaluate if a further adjuvant treatment with Trifluridine/Tipiracil could increase the rate of cases with undetectable ct-DNA and therefore improve DFS in a population at high-risk of relapse.

An additional target-driven cohort of HER2+ RAS wild-type colon cancer patients will be assessed for ct-DNA clearance after a tailored treatment with Trastuzumab and Tucatinib plus FOLFOX

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentre study, including two phase II randomized trials. In Part 1 resected stage III and high-risk stage II colon cancer patients with positive ct- DNA after surgery will be randomized to receive FOLFOX for 12 cycles or CAPOX for 8 cycles (at investigator choice) versus FOLFOXIRI for 12 cycles.

In Part 1 target-driven resected stage III and high-risk stage II HER2+ and RAS wild-type colon cancer patients with positive ct-DNA after surgery will receive Trastuzumab and Tucatinib plus FOLFOX for 12 cycles.

In Part 2 resected stage III and high-risk stage II colon cancer patients with positive ct- DNA after the end of a fluoropyrimidine and oxaliplatin-based adjuvant therapy - either in the frame or outside of Part 1 - will be randomized to receive observation or Trifluridine/Tipiracil for 6 cycles.

ELIGIBILITY:
Inclusion Criteria, Part I, adjuvant phase:

* Written informed consent to study procedures;
* 18 - 70 years of age ECOG Performance Status ≤ 1 or 71-75 years of age with ECOG Performance Status 0;
* Histologically confirmed stage III or high-risk stage II adenocarcinoma of colon including intraperitoneal rectal cancer. Stage II colon cancers are defined at high risk if at least one major prognostic factor (pT4, less than 12 nodes examined, clinical presentation with bowel perforation) or at least two minor prognostic factors (grade 3 or 4, clinical presentation with bowel obstruction, histological signs of vascular or lymphatic or perineural invasion, high preoperative CEA levels) are reported;
* Curative surgery performed no less than 4 and no more than 12 weeks prior to randomization (pending results of ct-DNA analysis, up to 2 cycles of FOLFOX/CAPOX are allowed to start the adjuvant treatment within 8-10 weeks after surgery);
* Contrast-enhanced chest and abdominal CT scan (or abdomen MRI and chest CT if contrast-enhanced CT scan is contraindicated) performed after the surgery and prior to randomization with no evidence of metastatic disease;
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue from the surgical specimen and blood sample for ct-DNA analysis within 28 days prior randomization;
* Positive ct-DNA after surgery (central assessment);
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥ 9 g/dl;
* Total bilirubin ≤1.5 fold the upper-normal limits (UNL), ASAT (SGOT) and/or ALAT (SGPT) ≤2.5 x UNL (or <5 x UNL in the case of liver metastases), alkaline phosphatase ≤2.5 x UNL (or <5 x UNL in case of liver metastases);
* Creatinine clearance ≥50 mL/min or serum creatinine ≤1.5 x UNL;
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For this trial, women of childbearing potential are defined as all women after puberty, unless the participants are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;
* Subjects and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception.

Contraception, starting during study screening visit throughout the study period up to 180 days after the last dose of chemotherapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;

- Will and ability to comply with the protocol.

Inclusion Criteria Part 1 and target-driven part 1, adjuvant phase II study

* Written informed consent to study procedures;
* 18 - 70 years of age ECOG PS ≤ 1 or 71-75 years of age with ECOG PS 0;
* Histologically confirmed stage III or high-risk stage II adenocarcinoma of colon including intraperitoneal rectal cancer. Stage II colon cancers are defined at high risk if at least one major prognostic factor (pT4, less than 12 nodes examined, clinical presentation with bowel perforation) or at least two minor prognostic factors (grade 3 or 4, clinical presentation with bowel obstruction, histological signs of vascular or lymphatic or perineural invasion, high preoperative CEA levels) are reported;
* For target-driven Part 1 only: HER2+ and RAS wt disease as determined by a tissue-based assay (central laboratory assessment);
* Curative surgery performed no less than 4 and no more than 12 weeks prior to randomization (pending results of ct-DNA analysis, up to 2 cycles of FOLFOX/CAPOX are allowed to start the adjuvant treatment within 8-10 weeks after surgery);
* Contrast-enhanced chest and abdominal CT scan (or abdomen MRI and chest CT if contrast-enhanced CT scan is contraindicated) performed after the surgery and prior to randomization with no evidence of metastatic disease;
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue from the surgical specimen and blood sample for ct-DNA analysis within 28 days prior randomization;
* Positive ct-DNA after surgery (central assessment);
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥ 9 g/dl;
* Total bilirubin ≤1.5 fold the upper-normal limits (UNL), ASAT (SGOT) and/or ALAT (SGPT) ≤2.5 x UNL, alkaline phosphatase ≤2.5 x UNL;
* Creatinine clearance ≥50 mL/min or serum creatinine ≤1.5 x UNL;
* For target-driven Part 1 only: Left ventricular ejection fraction (LVEF) ≥50% as assessed by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan.
* Availability of formalin-fixed, paraffin-embedded (FFPE) tumor tissue from the surgical specimen for translational analysis (only for patients eligible for protocol treatment);
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;
* Subjects and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception. Contraception, starting during study screening visit throughout the study period up to 180 days after the last dose of chemotherapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;
* Will and ability to comply with the protocol.

Inclusion Criteria, Part II, post-adjuvant phase:

* Written informed consent to study procedures;
* ≥ 18 years of age;
* Histologically confirmed stage III or high-risk stage II adenocarcinoma of colon including intraperitoneal rectal cancer. Stage II colon cancers are defined at high risk if at least one major prognostic factor (pT4, less than 12 nodes examined, clinical presentation with bowel perforation) or at least two minor prognostic factors (grade 3 or 4, clinical presentation with bowel obstruction, histological signs of vascular or lymphatic or perineural invasion, high preoperative CEA levels) are reported;
* Fluoropyrimidine and oxaliplatin-containing adjuvant treatment for at least 3 months (6 cycles of 5-fluorouracil and oxaliplatin-based therapy or 4 cycles of capecitabine and oxaliplatin-based-therapy) and no more than 6 months (12 cycles of 5-fluorouracil and oxaliplatin-based therapy or 8 cycles of capecitabine and oxaliplatin-based-therapy);
* Contrast-enhanced chest and abdominal CT scan (or abdomen MRI and chest CT if contrast-enhanced CT scan is contraindicated) performed within 4 weeks from the end of adjuvant therapy and 28 days prior to randomization;
* Availability of FFPE tumor tissue from the surgical specimen and blood sample for ct-DNA analysis within 28 days prior to randomization;
* Positive ct-DNA after the end of adjuvant treatment (centrally laboratory assessment);
* ECOG Performance Status ≤ 1;
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥9 g/dl;
* Total bilirubin ≤1.5 fold the upper-normal limits (UNL), ASAT (SGOT) and/or ALAT (SGPT) ≤2.5 x UNL (or <5 x UNL in the case of liver metastases), alkaline phosphatase ≤2.5 x UNL (or <5 x UNL in case of liver metastases);
* Creatinine clearance ≥ 50 mL/min or serum creatinine ≤1.5 x UNL;
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For this trial, women of childbearing potential are defined as all women after puberty, unless the participants are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;.
* Subjects and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception.

Contraception, starting during study screening visit throughout the study period up to 180 days after the last dose of chemotherapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;

- Will and ability to comply with the protocol.

Exclusion Criteria:

* Part 1, adjuvant phase and Part 2, post-adjuvant phase
* Any evidence of metastatic disease (radiological or pathological metastasis);
* Macroscopic or microscopic evidence of residual tumor (R1 or R2 resections) after surgery;
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ;
* For Part 1 only: patient with complete dihydropyrimidine dehydrogenase (DPYD) deficiency (homozygous of the following DPYD polymorphisms: c1679GG, c1905+1AA, c2846TT);
* History or evidence upon physical examination of CNS disease unless adequately treated;
* Clinical signs of malnutrition;
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating chemotherapy administration;
* Evidence of bleeding diathesis or coagulopathy;
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication;
* Significant vascular disease (i.e. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment;
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication;
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer);
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs;
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies;
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at screening. Sexually active males and females (of childbearing potential) unwilling to practice contraception (as defined in section 5.5) during the study and until 180 days after the last trial treatment.
* Part 1, target-driven, adjuvant phase:
* Ongoing ≥ Grade 2 diarrhea of any etiology at screening;
* Presence of known chronic liver disease;
* Known to be positive for hepatitis C infection (positive by polymerase chain reaction [PCR]). Subjects who have been treated for hepatitis C infection are permitted if they have documented sustained virologic response of at least 12 weeks.
* Known to be positive for hepatitis B (HBV) by surface antigen (HBsAg) expression. Subjects who are positive for either hepatitis B surface antibody (HBsAB) or antibodies to the hepatitis B core antigen (HBcAB) should be screened using PCR measurement of hepatitis B DNA levels. Subjects with hepatitis B DNA levels by PCR that require nucleoside analogue therapy are not eligible for the trial. The latest local guidelines should be followed regarding the monitoring of hepatitis B DNA levels by PCR subjects on study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
ct-DNA clearance rate after the end of the adjuvant treatment (ERASE-CRC part 1) | 6 months from the enrollment of the last patient in the adjuvant treatment
  Percentage of patients, relative to the total of enrolled subjects in the Part 1 of the study with undetectable ct-DNA at the end of adjuvant treatment.
ct-DNA clearance rate after the end of post-adjuvant treatment (ERASE-CRC part 2) | 6 months from the enrollment of the last patient in post-adjuvant treatment
  Percentage of patients, relative to the total of enrolled subjects in the Part 2 of the study with undetectable ct-DNA at the end of post-adjuvant treatment.
ct-DNA clearance rate after the end of target-driven adjuvant treatment (ERASE-CRC part 1 target-driven) | 6 months from the enrollment of the last patient in the target-driven adjuvant treatment
  Percentage of patients, relative to the total of enrolled subjects in the target-driven part
  1 of the study with undetectable ct-DNA at the end of adjuvant treatment.

SECONDARY OUTCOMES:
Overall Toxicity Rate 1 | 30 days from the last dose of the last patient in adjuvant treatment
  Percentage of patients, relative to the total of enrolled subjects in the Part 1 of the study, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during adjuvant treatment and follow-up.
Toxicity Rate 1 | 30 days from the last dose of the last patient in adjuvant treatment
  Percentage of patients, relative to the total of enrolled subjects in the Part 1 of the study, experiencing a specific adverse event of grade ≥ 3, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during adjuvant treatment and follow-up.
Disease Free Survival 1 (DFS1) | 60 months after the randomization of first patient in adjuvant treatment
  Time from randomization of the part 1 of the study to the first documentation of radiological disease relapse or death due to any cause, whichever occurs first. Secondary colorectal cancers are regarded as DFS events, whereas non-colorectal tumors are not. DFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of relapse for patients who are alive, on study and disease free at the time of the analysis. Alive patients having no tumor assessments after randomization will have time to event censored on the date of randomization.
Overall Survival 1 (OS1) | 60 months after the randomization of first patient in adjuvant treatment
  Time from randomization of the Part 1 of the study to the date of death due to any cause. For patients still alive at the time of the analysis, the OS time will be censored on the last date the patients were known to be alive.
Overall Toxicity Rate 2 | 30 days from the last dose of TRIFLURIDINE/TIPIRACIL
  Percentage of patients in the Part 2 of the study, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during post-adjuvant treatment and follow-up.
Toxicity Rate 2 | 30 days from the last dose of TRIFLURIDINE/TIPIRACIL
  Percentage of patients, relative to the total of enrolled subjects in the Part 2 of the study, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during postadjuvant treatment and follow-up.
Disease Free Survival 2 (DFS2) | 60 months after the randomization of first patient in post-adjuvant treatment
  Time from randomization of the part 2 of the study to the first radiological documentation of disease relapse or death due to any cause, whichever occurs first. Secondary colorectal cancers are regarded as DFS events, whereas non-colorectal tumors are not. DFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of relapse for patients who are alive, on study and disease free at the time of the analysis. Alive patients having no tumor assessments after randomization will have time to event censored on the date of randomization.
Overall Survival 2 (OS2) | 60 months after the randomization of first patient in post-adjuvant treatment
  Time from randomization of the part 2 of the study to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Overall Toxicity Rate TD1 | 30 days from the last dose of the last patient in target-driven adjuvant treatment
  Percentage of patients, relative to the total of enrolled subjects in the target-driven part 1 of the study, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during adjuvant treatment and follow-up.
Toxicity Rate TD1 | 30 days from the last dose of the last patient in target-driven adjuvant treatment
  percentage of patients, relative to the total of enrolled subjects in the target-driven part 1 of the study, experiencing a specific adverse event ≥ grade 3, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during adjuvant treatment and follow-up.
Disease Free Survival TD1 (DFS-TD1) | 60 months after the randomization of first patient in adjuvant treatment
  time from enrollment of the target-driven part 1 of the study to the first documentation of disease relapse or death due to any cause, whichever occurs first. Secondary colorectal cancers are regarded as DFS events, whereas non-colorectal tumors are not. DFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of relapse for patients who are alive, on study and disease free at the time of the analysis. Alive patients having no tumor assessments after enrollment will have time to event censored on the date of enrollment.
Overall survival TD1 (OS-TD1) | 60 months after the randomization of first patient in adjuvant treatment
  Time from enrollment of the target-driven part 1 of the study to the date of death due to any cause. For patients still alive at the time of the analysis, the OS time will be censored on the last date the patients were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Moretto, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (28):
- Italy (28):
  - Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Azienda Ospedaliera Cardinale Giovanni Panico, Tricase, Lecce
  - Ospedale San Donato di Arezzo, Arezzo
  - Spedali Civili di Brescia, Brescia
  - Fondazione POLIAMBULANZA ISTITUTO OSPEDALIERO, Brescia
  - AOU Cagliari PO Policlinico Universitario Duilio Casula Presidio Policlinico Universitario "Duilio Casula", Cagliari
  - A.O.U. di Ferrara Arcispedale Sant'Anna, Ferrara
  - A.O.U Careggi, Florence
  - E.O. Ospedali Galliera di Genova, Genova
  - Ospedale Misericordia di Grosseto, Grosseto
  - Azienda USL Toscana Nord Ovest di Livorno, Livorno
  - Ospedale San Luca di Lucca, Lucca
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - Fondazione IRCCS INT - Milano, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carita, Novara
  - Istituto Oncologico Veneto IOV - IRCCS, Padua
  - Azienda USL di Piacenza, Piacenza
  - Nuovo Ospedale di Prato, Prato
  - AUSL Romagna, Ravenna
  - Azienda USL IRCCS di Reggio Emilia (centro principale Reggio Emilia e centro satellite Guastalla)., Reggio Emilia
  - Policlinico Tor Vergata Roma, Roma
  - Istituto per la ricerca sui tumori Regina Elena, Roma
  - Policlinico Fondazione Agostino Gemelli, Roma
  - Ospedale Fatebenefratelli Isola Tiberina, Roma
  - Ospedale Campostaggia Poggiponsi, Siena
  - IRCCS di Candiolo, Torino
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine